CLINICAL TRIAL: NCT02849210
Title: A Phase I Multicenter, Open Clinical Trial With Subcutaneous Immunotherapy in Depot Presentation in Patients With Rhinoconjuncitivis Sensitized to Olea Europaea
Brief Title: A Clinical Trial With Subcutaneous Immunotherapy in Depot Presentation in Patients With Rhinoconjuncitivis Sensitized to Olea Europaea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-OLEA-DEPOT
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Rhinoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allergovac depot (Experimental): Allergovac depot with Olea europaea pollen extract
  Interventions: Biological: Allergovac depot with Olea europaea pollen extract

INTERVENTIONS:
Biological: Allergovac depot with Olea europaea pollen extract — Subcutaneous immunotherapy in depot presentation in a rapid dose escalation scheme: 6 weekly increasing dose injections at the initiation phase plus 3 maintenance monthly injections.

SUMMARY:
The study was designed according to the draft of allergenic product regulation published by Spanish Regulatory Agency. The aim of the study is to evaluate the safety and tolerability of subcutaneous immunotherapy with Olea europaea pollen extract in patients with rhinoconjunctivitis with or without associated mild asthma. In addition, surrogate efficacy parameters will be evaluated: immunoglobulin level changes and skin reactivity

DETAILED DESCRIPTION:
An study conducted througout Spain with 4000 allergic patients (Alergoloógica 2005) showed that 47% of patients with rhinoconjuncitivits and 51% of asthmatic patients were sentitized to olive pollen. This gives us an idea of the importance of this allergen sensitization in Spain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the informed consent form.
2. Patients must be between 18 and 60 years of age.
3. Patients with seasonal allergic rhinoconjunctivitis against Olea europea during a minimum of 2 years prior to study participation. Although allergic rhinoconjunctivitis is the pathology under study, the inclusion of patients with mild concomitant asthma is allowed.
4. Patients who obtained a prick test result ≥ 3 mm diameter to Olea europaea Positive and negative control of the test should give consistent results.
5. Patients with specific immunoglobulin E ≥ class 2 (CAP/PHADIA) to Olea europaea.
6. Patients sensitized to Olea europaea with clinically relevant symptoms in which treatment with Olea europea 100% vaccine is indicated.
7. Patients who met all windows of treatment described in the protocol for both, treatment and study procedures.
8. Women of childbearing potential must have a negative urine pregnancy test at Screening visit/Visit 0.
9. Women of childbearing potential must agree to use an appropriate contraception method during the study if they are sexually active.

Exclusion Criteria:

1. Patients who received immunotherapy in the previous 5 years for Olea europaea or for any allergen with cross reactivity or patients that are currently receiving immunotherapy for any allergen.
2. Patients with severe asthma or forzed expiratoy volumen in 1 second FEV1< 70% even if the are pharmacologically controlled .
3. Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator deems relevant so as to interfere with the study.
4. Polisensitized patients to other inhalant allergens besides Olea europaea, if in the judgment of the investigator may present symptoms clinically relevant to those other airborne allergens while participating in this study
5. Patients with a previous history of anaphylaxis
6. Patients with chronic urticaria,
7. Patients with moderate to severe atopic dermatitis
8. Patients who have participated in another clinical trial within 3 month prior to enrolment.
9. Patients under treatment with tricyclic antidepressives, phenothiazines , β-blockers, or Angiotensin Converting Enzyme Inhibitors (ACEI)
10. Female patients who are pregnant or breast-feeding
11. Patient who does not attend the visits
12. Patient's lack of collaboration or refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse reactions as a measure of Safety and tolerability | 17 weeks treatment period

SECONDARY OUTCOMES:
Immunoglobulin changes from baseline | At baseline and 1 week after last administered dose
Cutaneous reactivity changes from baseline | At baseline and 1 week after last administered dose
  Skin prick test will be conducted at baseline and 1 week after last administered dose to measure the wheal área changes in mm2

CONTACTS AND LOCATIONS:
Overall Officials: Maricruz Gómez Fernández, MD, Study Chair — Roxall Medicina España S.A
Locations (5):
- Spain (5):
  - Complejo Hospitalario de Jaén, Jaén, Andalusia
  - Hospital Santa Bárbara, Puertollano, Ciudad Real
  - Hospital Infanta Cristina, Badajoz
  - Hospital Costa de la Luz, Huelva
  - Hospital Nisar Sevilla, Seville